CLINICAL TRIAL: NCT02460757
Title: Glottic Width and Respiratory Flow in Patients With Various Lung Diseases
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Jane Winantea, Principal Investigator, University Hospital, Essen
Other Study IDs: RLKEssenVC
Record Dates: First submitted 2015-05-27; First posted 2015-06-02 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Lung Diseases
Keywords: glottic movement; emphysema; copd; vocal cord
MeSH Terms: conditions — Lung Diseases; Emphysema; Pulmonary Disease, Chronic Obstructive | interventions — Laryngoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with COPD
  Interventions: Other: Laryngoscopy
- Patients with interstitial lung disease
  Interventions: Other: Laryngoscopy
- Healthy subjects
  Interventions: Other: Laryngoscopy

INTERVENTIONS:
Other: Laryngoscopy — Observation of glottic width in different arms

SUMMARY:
In this study the investigators examine the glottic width and the respiratory flow at rest in patients with various lung disease. The investigators postulated that a positive expiratory pressure is created through the narrowing of the glottic width in patients with hyperinflation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for a bronchoscopy
* Minimum age of 18 years
* Signed informed consent

Exclusion Criteria:

* Patients requiring mechanical ventilation during bronchoscopy
* Disease of the larynx
* Inability to breathe through the mouthpiece

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with various lung diseases in a primary care clinic
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Angle of the glottic width | 18 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Ruhrlandklinik, Essen, Germany